CLINICAL TRIAL: NCT00968136
Title: Short-term Ketogenic Diet as Compared With Conventional Long-term Trial in Refractory Infantile Spasms: A Randomized, Controlled Study
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Other Study IDs: 4-2006-0020
Record Dates: First submitted 2009-08-27; First posted 2009-08-28 (Estimated); Last update posted 2009-08-28 (Estimated); Status verified 2009-08

CONDITIONS: Infantile Spasms
Keywords: refractory infantile spasms
MeSH Terms: conditions — Spasms, Infantile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- a short-term trial of the ketogenic diet
- long-term trial of the ketogenic diet.

SUMMARY:
This is a randomized, controlled study to compare Short-term ketogenic diet with conventional long-term trial in refractory infantile spasms.

ELIGIBILITY:
Inclusion Criteria:

1. Patients, who have recalcitrant infantile spasms and undertake the ketogenic diet at Severance Hospital and Sanggye Paik Hospital from 2005 to 2008.
2. Clinical and electroencephalography findings are compatible with infantile spasms
3. Spasms are intractable to the initial combination of vigabatrin (150 mg/kg) and topiramate (10 mg/kg) and/or additional indicated anti-epileptic drugs including prednisolone (2 mg/kg for 2 weeks and an additional 2 weeks for tapering).
4. Study entry requires magnetic resonance imaging to confirm the absence of a progressive cerebral lesion.

Exclusion Criteria:

1. Patients who have a history of hyperlipidaemia and underlying metabolic diseases including acute intermittent porphyria, pyruvate carboxylase deficiency, and fatty acid oxidation defects.
2. Patients who have a history of nephrolithiasis.

Ages: 1 Month to 5 Years | Sex: All
Age Groups: Child
Study Population: refractory infantile spasms
Sampling Method: Non-Probability Sample

PRIMARY OUTCOMES:
Primary outcome measures include seizure relapse and frequency after successful completion of the ketogenic diet. | Finally, 35 patients could be followed up for more than 12 months after successful discontinuation of the diet and then primary outcome will be measured.